CLINICAL TRIAL: NCT03990402
Title: GHR (Global Health Research) Project:17/63/38 - NIHR (National Institute for Health Research) Global Health Research Group on Improving Asthma Outcomes in African Children at Queen Mary University of London
Brief Title: Achieving Control of Asthma in Children In Africa
Acronym: ACACIA
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Jonathan Grigg, Professor of Paediatric Respiratory and Environmental Medicine, Queen Mary University of London
Other Study IDs: 269211
Record Dates: First submitted 2019-01-08; First posted 2019-06-19 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Asthma
Keywords: FeNO; Africa; Spirometry; Asthma Control; ACT; Prevalence
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Malawi group: 500 young people with asthma symptoms in Malawi
- South Africa group: 500 young people with asthma symptoms in South Africa
- Uganda group: 500 young people with asthma symptoms in Uganda
- Nigeria: 500 young people with asthma symptoms in Nigeria
- Zimbabwe group: 500 young people with asthma symptoms in Zimbabwe
- Ghana group: 500 young people with asthma symptoms in Ghana

SUMMARY:
The main aim of the study is to identify altogether 3000 children aged between 12 and 16 years old with asthma symptoms in six sub-Saharan African countries. The study furthermore aims to assess their asthma control, current treatment, knowledge of and attitudes to asthma, as well as the barriers to achieving good asthma control.

DETAILED DESCRIPTION:
Asthma prevalence in young people has been rising in several African countries during the last decade, reaching between 10% and 20% in Central Africa, and up to 20% in South Africa. In addition, asthma related mortality in many African countries is high. South Africa has the third highest asthma related mortality rate in the world. Yet to date, a lack of asthma research and research infrastructure means that we do not have the evidence to either inform advocacy or to develop interventions that improve asthma outcomes.

This study aims to collect data about asthma prevalence and to identify existing barriers to effective asthma management of young people in 6 sub-Saharan countries: Malawi, South Africa, Zimbabwe, Uganda, Ghana, and Nigeria. Each of these countries identifies 500 young people with asthma between 12 and 16 years of age through a screening questionnaire in schools. These 3000 young people with asthma symptoms fill in a survey about asthma, including questions around asthma control, current treatment and access to care, asthma knowledge, asthma attitudes, smoking and environmental influences. Some of the participants also discuss asthma related topics in focus groups. A subset of the participants furthermore do Spirometry and FeNO testing. In addition to the data collection, the study develops and tests options for an intervention aimed at improving asthma control, including the adaption of a United Kingdom - based theater play about asthma awareness. The development of WiFi infrastructure and IT solutions is promoted by the study, where appropriate.

ELIGIBILITY:
Inclusion Criteria:

* aged between a minimum of 12 years, and
* a maximum of 14 years

Exclusion Criteria:

* Age less than 12 years
* age more than 14 years

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Young people between 12 and 14 years of age.
Sampling Method: Probability Sample
Enrollment: 3767 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of children with asthma symptoms or asthma | 12 months
  Percentage of children with asthma or asthma symptoms, based on GAN (Global Asthma Network) screening tool.

SECONDARY OUTCOMES:
Understanding about Asthma - Questions | 1 year
  set of questions about asthma knowledge, maximum knowledge score is 13, minimum knowledge score is 0, total range is 13. Higher values represent better knowledge.
Brief Illness Perception Questionnaire | 1 year
  Each of the 9 items in the Brief Illness Perception Questionnaire has a minimum score of 0 and a maximum score of 10.
  The consequences score is the response to item 1. The timeline score is the response to item 2. The personal control scores is the response to item 3. The treatment control score is the response to item 4. The identity score is the response to item 5. The coherence score is the response to item 7. The emotional representation is the response to item 8. Illness concern is measured by item 6. Item 9 is the causal item.
  Overall score which represents the degree to which the illness is perceived as threatening or benign. To compute that score, reverse score items 3, 4, and 7 and add these to items 1, 2, 5, 6, and 8. A higher score reflects a more threatening view of the illness. The overall score has a minimum score of 0 and a maximum score is 80.
Asthma control test | 4 weeks
  using validated ACT - Asthma Control Test (license by GlaxoSmithKlyne). The minimum score is 5 (poor control of asthma), the maximum score is 25 (complete control of asthma). An ACT score >19 indicates well-controlled asthma
environmental factor assessment | 1 year
  questions related to the environment of young people with asthma symptoms, reported using descriptive statistics, and percentages
access to medical care of young people with asthma | 1 year
  set of questions related to access to medical care, reported using descriptive statistics, and percentages
current treatment of asthma | 1 year
  set of questions about current medication, reported using descriptive statistics, and percentages
Adherence to medication | 1 year
  set of questions asking about adherence to medication, reported as descriptive statistics and percentages, as well as free text comments.
asthma-related time off school | 4 weeks
  questions asking about asthma-related time off school, reported as descriptive statistics and percentages
smoking | 1 year
  questions assessing active and passive smoking, reported as descriptive statistics and percentages
FeNO (fractional exhaled nitric oxide) | up to 1 day
  FeNO measurements - exhaled Nitric Oxide
Spirometry FEV1 | up to 1 day
  FEV1, in liter, and in liter predicted
Asthma Control according to GINA (Global INitiative for Asthma) | 4 weeks
  GINA questionnaire (Global INitiative for Asthma) using four questions, assessing control of asthma symptoms. Outcome is 'well controlled' if none of the four questions is answered 'Yes', 'partly controlled' if one or two of the four questions is answered 'Yes', uncontrolled, if three or four of the four questions is answered 'Yes'.
Spirometry FVC | up to 1 day
  FVC, in liter, and in liter predicted
Spirometry FEV1/FVC | up to 1 day
  Ratio of FEV1 to FVC
FEF25-75 | up to 1 day
  FEF25-75 as percentage

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Grigg, Professor, Principal Investigator — Queen Mary University of London, Blizard Institute
Locations (6):
- Kwame Nkrumah University of Science & Technology (KNUST), Kumasi, Ashanti Region, Ghana
- Malawi-Liverpool-Wellcome Trust Clinical Research Programme, Blantyre, Malawi
- Lagos State University College of Medicine, Lagos, Nigeria
- University of Kwa-Zulu Natal, Durban, KwaZulu-Natal, South Africa
- Makarere University College of Health Sciences, Kampala, Uganda
- University of Zimbabwe College of Health Sciences, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Undecided
We are currently working on a detailed plan to share the collected data with other researchers in accordance with the existing data protection legislation.

REFERENCES:
- [Derived] Oyenuga VO, Mosler G, Addo-Yobo E, Adeyeye OO, Arhin B, Fortune F, Griffiths CJ, Kasekete M, Mkutumula E, Mphahlele R, Mujuru HA, Muyemayema S, Nantanda R, Nkhalamba LM, Ojo OT, Owusu SK, Ticklay I, Ubuane PO, Yakubu RC, Zurba L, Masekela R, Grigg J. Asthma symptoms, severity, and control with and without a clinical diagnosis of asthma in early adolescence in sub-Saharan Africa: a multi-country, school-based, cross-sectional study. Lancet Child Adolesc Health. 2024 Dec;8(12):859-871. doi: 10.1016/S2352-4642(24)00232-3. Epub 2024 Oct 21. PMID 39447587